CLINICAL TRIAL: NCT07052474
Title: Intensive Trauma-Focused Treatment for Adolescents With Post-Traumatic Stress Disorder (PTSD): Feasibility and Preliminary Effects
Brief Title: Intensive Trauma-Focused Treatment for Adolescents With PTSD: Feasibility and Preliminary Effects
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Helander, PhD, Licenced psychologist, Karolinska Institutet
Other Study IDs: DNR2023-06501-01
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; Intensive treatment; Adolescents; Brief Intensive Trauma Treatment
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PTSD referred to the trauma unit at Child- and adolescent psychiatry, Stockholm: Patients included in the study receive one week of intensive trauma-focused treatment where two different evidence-based treatments are combined with physical activity and family support.
  Interventions: Behavioral: Intensive trauma-focused treatment

INTERVENTIONS:
Behavioral: Intensive trauma-focused treatment — The treatment program includes components of Trauma focused cognitive behavioral therapy (TF-CBT), Eye Movement Desensitization and Reprocessing Therapy (EMDR), physical activity, as well as parent sessions. The intensive treatment largely follows the Dutch intensive trauma treatment program "Korte Intensieve Traumabehandeling" (KIT) (Albisser et al., 2024).
  The intensive treatment incorporates core components from TF-CBT for children and adolescents (Cohen & Mannarino, 2008) as well as the standard EMDR protocol (Shapiro, 2018).

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) in adolescents is a debilitating condition that, without timely intervention, risks becoming chronic and severely impairing development. Although evidence-based treatments such as Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) and Eye Movement Desensitization and Reprocessing (EMDR) are effective, they typically require weekly sessions over 6-9 months, which many adolescents struggle to complete. High dropout rates remain a significant clinical challenge.

Intensive trauma-focused interventions have shown promising outcomes in adults, including rapid symptom reduction and improved retention. Inspired by a Dutch model, this project evaluates a Swedish adaptation of Korte Intensieve Traumabehandeling (KIT), which combines EMDR, elements of TF-CBT, physical activity, and parental support in a 5-day intensive treatment.

This project is a pilot study to examine the feasibility, early effects, and practicality of intensive trauma-focused therapy. The pilot study is the first step toward planning a larger, controlled study in Swedish child and adolescent psychiatry.

The following questions are included in the project:

1. Is intensive trauma-focused psychological treatment with EMDR, components of TF-CBT, combined with physical activity and a parent group a feasible, suitable, and acceptable treatment method for PTSD within Swedish child and adolescent psychiatry in terms of:

   1. Therapists' ratings of whether they find the intensive trauma-focused treatment acceptable, appropriate, and feasible.
   2. The number of patients who complete the treatment without dropping out
   3. Patients' self-reported satisfaction with the treatment
   4. The proportion of patients with "adverse effects"
2. Does intensive trauma-focused psychological treatment with EMDR, components of TF-CBT, combined with physical activity and a parent group for PTSD, lead to a decrease in symptoms in the expected direction in terms of:

   1. PTSD symptoms
   2. General mental health

DETAILED DESCRIPTION:
Background Post-Traumatic Stress Disorder (PTSD) is associated with a high risk of chronicity if untreated. Rapid and effective interventions are crucial for reducing symptom burden and preventing long-term complications. According to NICE treatment guidelines, the two primary recommended treatments for PTSD in children and adolescents are Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) and Eye Movement Desensitization and Reprocessing (EMDR), both of which are supported by substantial empirical evidence. These treatments typically involve 6-9 months of weekly sessions.

A notable challenge in treating adolescents with PTSD is the high rate of premature treatment termination. Increasing treatment intensity may reduce dropout rates, as studies indicate that more frequent sessions lead to greater symptom reduction and improved retention. In adult populations, intensive programs that combine evidence-based therapies such as EMDR and Prolonged Exposure (PE), alongside physical activity and psychoeducation, have shown promising results, including significant symptom reduction and lower dropout rates.

While EMDR and exposure-based therapies share some similarities, they operate through different mechanisms. TF-CBT utilizes continuous exposure to facilitate habituation and fear extinction, whereas EMDR employs dual attention stimulation, often via eye movements. The hypothesis that combining both approaches can enhance treatment effects through complementary mechanisms requires further investigation, particularly in an intensive format.

For adolescents, treatment protocols similar to those developed for adults have emerged, evaluating variations of 5-8 days of intensive treatment that integrate therapeutic modalities such as EMDR and CBT-based treatments like PE or TF-CBT, along with parental support and physical activity. In the Netherlands, a Brief Intensive Trauma Treatment (KIT; Korte Intensieve Traumabehandeling) model has been developed, which combines EMDR with TF-CBT, physical exercise, and parental support.

Despite promising outcomes indicating rapid symptom alleviation-often within a week-existing research on intensive trauma treatments for children and adolescents is limited. Notably, no randomized controlled trials (RCTs) have been published, and many studies lack control groups. Observed results suggest that the majority of participants no longer meet PTSD diagnostic criteria post-treatment while reporting reduced depressive symptoms. However, methodological limitations call for cautious interpretation of these findings.

This project is designed as a feasibility study utilizing a within-group design to assess the viability and preliminary effects of a Swedish adaptation of the KIT model. This intensive five-day trauma-focused intervention will incorporate EMDR and TF-CBT elements alongside physical activity and parent sessions, targeting adolescents with PTSD referred to the Child and Adolescent Psychiatry (CAP) Trauma Unit in Stockholm. Ethical approval for the study has been granted (Dnr 2024-05726-02).

Time points for data assessment Data is collected at baseline and at five weeks post treatment week for all measures. In addition, two of the measures are collected with higher intensity, the CRIES 13, self rated measure of PTSD symptoms is collected daily during the treatment week and at one and two weeks post treatment. The CATS 2 is assessed at one and two weeks post treatment by both the patient and the caregiver.

Data Analysis As a pilot study with a limited sample size, inferential statistics are not planned. Instead, changes in PTSD symptoms and mental health will be examined descriptively. Planned analyses include within-group effect sizes, proportion of treatment drop-out, and proportions of patients in full or partial remission. Attrition rates will be compared to dropout rates reported in earlier studies.

ELIGIBILITY:
Patients with PTSD between 13 and 17 years of age who are referred to the specialized trauma unit within Stockholm Child and Adolescent Psychiatry. Patients who meet inclusion criteria after assessment at the BUP Trauma Unit are informed about the study. If interested, they attend a meeting to receive further information and provide consent. Background data is collected, and a diagnostic interview (CAPS-CA-5) is scheduled. Inclusion is decided during treatment planning meetings.

Inclusion Criteria:

* Diagnosis of PTSD
* No or stable medication involving antidepressants, stimulants, and/or antipsychotics
* At least one caregiver can participate in the treatment

Exclusion Criteria:

* High risk for suicide
* IQ below 75
* Current substance abuse

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients referred to the CAP Stockholm Trauma unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), och Feasibility of Intervention Measure (FIM). | From treatment start to five weeks after the intensive treatment week.
  The therapist rated measures of how acceptable, appropriate, and feasible the treatment is perceived. The measures consist of three scales with four items each and have demonstrated strong psychometric properties. Items are rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Minimum value 4, maximum value 20. A higher value indicates a better outcome.
  To consider the intervention acceptable, appropriate, and feasible, at least 80% of clinicians must rate the method above 50 on a 0-100 scale on the AIM, IAM, and FIM subscales.

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 - Child/Adolescent Version (CAPS-CA-5) | Assessment before treatment start and five weeks after treatment week.
  The CAPS-CA-5 is a structured diagnostic interview assessing PTSD diagnosis. It contains 30 items and assesses symptom severity by combining frequency and intensity ratings on a 0-4 scale, minimum value = 0, maximum value = 120
  CAPS-CA-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Similarly, CAPS-CA-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). PTSD diagnostic status is determined by first dichotomizing each symptom as "present" or "absent," then following the DSM-5 diagnostic rule. A symptom is considered present only if the corresponding item severity score is rated 2 ("moderate/threshold") or higher.
The Children Impact of Event Scale | Before treatment, every day during the five-day intensive treatment, and at one, two, four, and five weeks post the treatment week.
  CRIES-13 is a 13-item scale assessing PTSD symptoms using a four-point Likert scale (Not at all, Rarely, Sometimes, Often), scored 0,1,3,5 with no reversed items. It includes subscales for intrusion (four items), avoidance (four items), and arousal (five items). The total score thus ranges from 0 to 65 on this 13-item scale. A higher score indicates a worse outcome in terms of PTSD symptom burden.
Child and adolescent trauma screen 2 | Pre treatment, one, two, four and five weeks post the treatment week
  Trauma symptoms are assessed using the CATS-2, both for the adolescent (CATS-2-U) and for the caregiver (CATS-2-F). This trauma questionnaire screens for both trauma history and trauma symptoms based on DSM-5 criteria. The CATS-2 consists of two parts. Part one is a screening for potentially traumatic events at any point in the individual's life, comprising 15 items where the patient can answer YES or NO. Part two is a screening for post-traumatic symptoms over the past four weeks, with 20 items and five questions about how the child's daily life has been impacted by these symptoms. The total score for CATS-2-U may vary between 0 and 60 points. Each item is rated on a four-point Likert scale between 0 (never) to 3 (almost always), and the total score is calculated by summing the answers from each item. A higher score indicates a worse outcome.
Strengths and Difficulties Questionnaire | Assessment before treatment and at five weeks follow-up.
  The Strengths and Difficulties Questionnaire is a 25-item scale assessing general psychological functioning. A total difficulties score is generated by summing scores from all the scales except the prosocial scale, with a minimum value of 0 to a maximum value of 40. Each subscale consists of 5 items each (range 0-2 from "not true", to "certainly true". A higher score indicates a worse outcome.
Client Satisfactory Questionnaire-8 (CSQ-8) | Assessed at five weeks follow-up.
  The Client Satisfaction Questionnaire-8 is an 8-item self-report scale measuring satisfaction with treatment. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

OTHER OUTCOMES:
Adverse effects checklist | Daily during the treatment period and at one, two, four and five weeks post treatment week
  The patients are asked if she/he has self-harmed, had suicidal thoughts and/or if he/she has had sought for akute psychiatric treatment
Drop out of treatment | Any treatment dropout during the five-day treatment period.
  The proportion of patients that has dropped out of treatment is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helander, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Centre for Psychiatry Research, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD was not included in the ethical permission.

REFERENCES:
- [Background] Pynoos, R. S., Weathers, F. W., Steinberg, A. M., Marx, B. P., Layne, C. M., Kaloupek, D. G., ... & Kriegler, J. A. (2015). Clinician-administered PTSD scale for DSM-5-child/adolescent version. Scale available from the National Center for PTSD at www. ptsd. va. gov.
- [Background] Mevissen L, Ooms-Evers M, Serra M, de Jongh A, Didden R. Feasibility and potential effectiveness of an intensive trauma-focused treatment programme for families with PTSD and mild intellectual disability. Eur J Psychotraumatol. 2020 Jul 14;11(1):1777809. doi: 10.1080/20008198.2020.1777809. PMID 33029319
- [Background] Hendriks L, de Kleine RA, Heyvaert M, Becker ES, Hendriks GJ, van Minnen A. Intensive prolonged exposure treatment for adolescent complex posttraumatic stress disorder: a single-trial design. J Child Psychol Psychiatry. 2017 Nov;58(11):1229-1238. doi: 10.1111/jcpp.12756. Epub 2017 Jun 14. PMID 29057522
- [Background] Ooms-Evers M, van der Graaf-Loman S, van Duijvenbode N, Mevissen L, Didden R. Intensive clinical trauma treatment for children and adolescents with mild intellectual disability or borderline intellectual functioning: A pilot study. Res Dev Disabil. 2021 Oct;117:104030. doi: 10.1016/j.ridd.2021.104030. Epub 2021 Jul 24. PMID 34314951
- [Background] Wachen, J. S., Dondanville, K. A., Evans, W. R., Morris, K., & Cole, A. (2019). Adjusting the Timeframe of Evidence-Based Therapies for PTSD-Massed Treatments. In Current Treatment Options in Psychiatry (Vol. 6, Issue 2, pp. 107-118). Springer. https://doi.org/10.1007/s40501-019-00169-9
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Dyregrov A, Kuterovac G, Barath A. Factor analysis of the impact of event scale with children in war. Scand J Psychol. 1996 Dec;37(4):339-50. doi: 10.1111/j.1467-9450.1996.tb00667.x. PMID 8931390
- [Background] Nader, K., Kriegler, K. A., Blake, D. D., Pynoos, R. S., Newman, E., & Weathers, F. W. (1996). Clinician-administered PTSD scale for children and adolescents.
- [Background] Sachser C, Berliner L, Risch E, Rosner R, Birkeland MS, Eilers R, Hafstad GS, Pfeiffer E, Plener PL, Jensen TK. The child and Adolescent Trauma Screen 2 (CATS-2) - validation of an instrument to measure DSM-5 and ICD-11 PTSD and complex PTSD in children and adolescents. Eur J Psychotraumatol. 2022 Aug 1;13(2):2105580. doi: 10.1080/20008066.2022.2105580. eCollection 2022. PMID 35928521
- [Background] Van Woudenberg C, Voorendonk EM, Bongaerts H, Zoet HA, Verhagen M, Lee CW, van Minnen A, De Jongh A. Effectiveness of an intensive treatment programme combining prolonged exposure and eye movement desensitization and reprocessing for severe post-traumatic stress disorder. Eur J Psychotraumatol. 2018 Jul 10;9(1):1487225. doi: 10.1080/20008198.2018.1487225. eCollection 2018. PMID 30013726
- [Background] van Pelt Y, Fokkema P, de Roos C, de Jongh A. Effectiveness of an intensive treatment programme combining prolonged exposure and EMDR therapy for adolescents suffering from severe post-traumatic stress disorder. Eur J Psychotraumatol. 2021 May 14;12(1):1917876. doi: 10.1080/20008198.2021.1917876. PMID 34025927
- [Background] Van Minnen A, Voorendonk EM, Rozendaal L, de Jongh A. Sequence matters: Combining Prolonged Exposure and EMDR therapy for PTSD. Psychiatry Res. 2020 Aug;290:113032. doi: 10.1016/j.psychres.2020.113032. Epub 2020 May 16. PMID 32454314
- [Background] Tinghog P, Vagbratt L, Jennstal J, Bragesjo M, Moller N. Acceptability and Preliminary Effects of Intensive Brief Trauma-Focused PTSD Treatment for Refugees. Torture. 2024;34(3):54-63. doi: 10.7146/torture.v34i3.147953. PMID 39878600
- [Background] Simmons C, Meiser-Stedman R, Baily H, Beazley P. A meta-analysis of dropout from evidence-based psychological treatment for post-traumatic stress disorder (PTSD) in children and young people. Eur J Psychotraumatol. 2021 Aug 5;12(1):1947570. doi: 10.1080/20008198.2021.1947570. eCollection 2021. PMID 34377359
- [Background] Shapiro, F. (2007). EMDR, Adaptive Information Processing, and Case Conceptualization. Journal of EMDR Practice and Research, 1(2), 68-87. https://doi.org/10.1891/1933-3196.1.2.68
- [Background] John-Baptiste Bastien R, Jongsma HE, Kabadayi M, Billings J. The effectiveness of psychological interventions for post-traumatic stress disorder in children, adolescents and young adults: a systematic review and meta-analysis. Psychol Med. 2020 Jul;50(10):1598-1612. doi: 10.1017/S0033291720002007. Epub 2020 Jun 22. PMID 32624017
- [Background] Post-traumatic stress disorder NICE guideline. (2018). www.nice.org.uk/guidance/ng116
- [Background] Pietrzak RH, Goldstein RB, Southwick SM, Grant BF. Psychiatric comorbidity of full and partial posttraumatic stress disorder among older adults in the United States: results from wave 2 of the National Epidemiologic Survey on Alcohol and Related Conditions. Am J Geriatr Psychiatry. 2012 May;20(5):380-90. doi: 10.1097/JGP.0b013e31820d92e7. PMID 22522959
- [Background] Cohen JA, Deblinger E, Mannarino AP. Trauma-focused cognitive behavioral therapy for children and families. Psychother Res. 2018 Jan;28(1):47-57. doi: 10.1080/10503307.2016.1208375. Epub 2016 Jul 22. PMID 27449400
- [Background] Albisser, N., Westerveld, M., Kooij, L., de Keizer-Altink, M., & Lindauer, R. (2024). Korte intensieve traumabehandeling bij jongeren. Kind & Adolescent Praktijk, 23(3), 16-24. https://doi.org/10.1007/s12454-024-1833-1
- See also: Related Info — https://ki.se/en/cns/research/centre-for-psychiatry-research

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT07052474/Prot_SAP_000.pdf